CLINICAL TRIAL: NCT00297050
Title: A Phase I Double-Blind, Placebo-Controlled, Dose-Escalating Study to Evaluate the Safety and Tolerability of Intravenous Peramivir in Healthy Subjects
Brief Title: Safety and Dose Study of Peramivir for Influenza Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060105; 06-I-0105
Record Dates: First submitted 2006-02-25; First posted 2006-02-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-08-05

CONDITIONS: Influenza
Keywords: Influenza Virus; Avian Influenza; Normal Volunteers; Neuraminidase Inhibitor; Viral Disease; Healthy Volunteer; HV
MeSH Terms: conditions — Influenza, Human; Influenza in Birds; Virus Diseases | interventions — peramivir

INTERVENTIONS:
Drug: Peramivir

SUMMARY:
This study will evaluate the safety and tolerability of peramivir, a new drug to treat influenza. The study will administer gradually increasing doses of the drug in successive small groups of subjects to determine the optimal dose that is safe and well tolerated. It will be studied first at a single dose and then in multiple doses. The study will also determine how long peramivir stays in the body and how high the drug levels are in the blood.

Men and women 18 - 40 years of age who weigh at least 110 lbs. and have a body mass index (BMI) between 19 and 32 may be eligible for this study. Candidates are screened with a medical history, physical examination, electrocardiogram (EKG), and blood and urine tests.

Part I - Single Dose Escalation

Participants are admitted to the NIH hospital for 32 to 40 hours for a single 15-minute intravenous infusion of peramivir or placebo (saline), followed by monitoring and evaluation. The drug dose is increased in successive groups of eight subjects; in each group, six subjects are given peramivir and two receive placebo. The first group receives 0.5 mg/kg of peramivir; subsequent groups receive increasingly higher doses (1, 2, 3.5, and 5 mg/kg) as long as the last dose was well tolerated by the preceding group. Blood samples are drawn and subjects are monitored for vital signs (temperature, blood pressure and heart rate) and for symptoms such as headache, nausea, shortness of breath or pain at 0.5, 1, 2, 3, 6, 9, 12, 18 and 24 hours after the drug infusion. At the 24-hour evaluation they have an EKG. If needed, an echocardiogram (ultrasound examination of the heart) may also be done. Subjects return to the clinic 2, 3, 7, 14, and 28 days after the infusion for a check of vital signs, review of symptoms, blood draw, and urine sample collection. In addition, subjects are asked to collect all their urine for the first 48 hours after the study drug infusion.

Part II - Multi-dose Escalation

Groups of 16 subjects receive an intravenous infusion of peramivir (12 subject) or placebo (4 subjects) once a day for 5 consecutive days. The first four infusions are given in the NIH outpatient clinic. The dose of peramivir is increased in successive groups of 16 subjects as long as the preceding dose was well tolerated. Before the infusion on day 1, subjects have a physical examination, blood test and EKG to obtain baseline values. After the infusion, they remain in the hospital for 6 hours. Vital signs and symptoms are c...

DETAILED DESCRIPTION:
Human influenza is a serious disease causing over 30,000 deaths in the United States each year, and avian influenza presents a threat of a future pandemic. Despite this burden of current and potential disease, there are no parenteral treatments for influenza, and currently, the most common treatment (oseltamivir) is expensive and complex to manufacture.

The primary purpose of this protocol is to evaluate the safety and tolerability of intravenous peramivir, a neuraminidase inhibitor. Beginning with a low single-dose, the safety and tolerability is established by evaluating symptoms, clinical laboratory tests, ECG, and pharmacokinetics. Utilizing a series of stopping rules and a medical monitor, the dose will be escalated as safety and tolerability are established. Once the maximum tolerated dose (MTD) is established in the first part of this trial (either limited by adverse effects or up to maximum anticipated dose), the safety and tolerability of multi-dose administration will begin (replicating anticipated clinical use). These cohorts will be evaluated using similar criteria. The dose used in the multi-dose cohorts will also be escalated as safety and tolerability are established.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age greater than or equal to 18 years and less than or equal to 50 years.
  2. Weight greater than or equal to 50 kg (110 lbs).
  3. Body mass index (BMI) of 19-32 kg/m(2).
  4. Subjects must agree to:
* Not take any prescription or OTC medications with the exception of Tylenol, and contraceptive medications for a period of 7 days prior and during study drug administration.
* Not consume any alcohol for a period of 2 days prior and during study drug administration.
* Not receive a live attenuated influenza vaccine (Flumist) for 7 days prior to study drug administration, through day 14 (which will be at least 8 days from the last dose of study drug).
* Not participate in any other research protocol between screening, and the last day of follow-up.

  5. Females of child-bearing potential must (one of the following):
* Be surgically sterile.
* Be abstinent (or willing to be) 4 weeks prior to date of screening evaluation through 4 weeks after study drug administration.
* Use oral contraceptives, or other form of hormonal birth control including hormonal vaginal rings or transdermal patches, and have been using these for three months prior through 4 weeks after study drug administration.
* Use an intra-uterine device (IUD) as birth control 4 weeks prior to date of screening evaluation through 4 weeks after study drug administration.
* Use (by ensuring her male partner(s) uses) barrier contraception (condom) with a spermacide as birth control 4 weeks prior to date of screening evaluation through 4 weeks after study drug administration.

EXCLUSION CRITERIA:

1. Any chronic medical problem that requires daily oral medications (except Tylenol and oral contraceptives), or other medical history that in the opinion of the investigator significantly increases the risk associated with a Phase I drug.
2. History of cardiovascular disease or unexplained syncope
3. Family history of sudden death in a first degree relative.
4. Women who are breast-feeding.
5. Positive urine or serum pregnancy test.
6. Abnormal ECG (defined as any baseline Grade 1 or greater toxicity by the toxicity table for ECG. The toxicity table specifically evaluates PR interval, QTc interval and rhythm. Asymptomatic sinus bradycardia, especially in a subject that exercises, is acceptable).
7. Abnormal chemistry panel (defined as any baseline Grade 1 or greater toxicity from the Chem 20 panel evaluating only sodium, potassium, total CO2 (bicarbonate), creatinine, glucose, urea nitrogen, total calcium, total magnesium, phosphorus, alkaline phosphatase, ALT, AST, total bilirubin, direct bilirubin, LDH, total protein, total CK, uric acid).
8. Abnormal complete blood count (CBC) (defined as any baseline Grade 1 or greater toxicity from the CBC evaluating only the WBC, hemoglobin, hematocrit, and platelets).
9. Abnormal urinalysis (defined as any baseline Grade 1 or greater toxicity from the urinalysis evaluating only protein, and RBCs).
10. Positive serology for Hepatitis B surface antigen.
11. Positive serology for Hepatitis C.
12. Positive serology for HIV-1.
13. Positive urine drug screen.
14. Participation in a study of any investigational drug within the last 30 days.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100
Dates: Start 2006-02-23; Primary Completion 2006-11-14 (Actual); Study Completion 2006-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cox NJ, Subbarao K. Influenza. Lancet. 1999 Oct 9;354(9186):1277-82. doi: 10.1016/S0140-6736(99)01241-6. PMID 10520648
- [Background] Thompson WW, Shay DK, Weintraub E, Brammer L, Cox N, Anderson LJ, Fukuda K. Mortality associated with influenza and respiratory syncytial virus in the United States. JAMA. 2003 Jan 8;289(2):179-86. doi: 10.1001/jama.289.2.179. PMID 12517228
- [Background] Beigel JH, Farrar J, Han AM, Hayden FG, Hyer R, de Jong MD, Lochindarat S, Nguyen TK, Nguyen TH, Tran TH, Nicoll A, Touch S, Yuen KY; Writing Committee of the World Health Organization (WHO) Consultation on Human Influenza A/H5. Avian influenza A (H5N1) infection in humans. N Engl J Med. 2005 Sep 29;353(13):1374-85. doi: 10.1056/NEJMra052211. No abstract available. PMID 16192482